CLINICAL TRIAL: NCT03246789
Title: Reaching and Engaging Depressed Senior Center Clients
Brief Title: Reaching and Engaging Depressed Senior Center Clients (REDS)
Acronym: REDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York City Department for the Aging (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1704018114; P50MH113838 (NIH)
Record Dates: First submitted 2017-08-03; First posted 2017-08-11 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-02

CONDITIONS: Depression, Unipolar; Mental Health Disorder
MeSH Terms: conditions — Depressive Disorder; Mental Disorders | interventions — Health

STUDY DESIGN:
Intervention Model Description: Investigators will randomly assign four senior centers to offer either Engage-M (N=40), the treatment offered by REDS (1 individual and 8 weekly group sessions) or 8 group sessions "Wellness in Mind and Body" plus mental health referral (W-MH; N=20). Participants will have clinically significant depressive symptoms (PHQ-9>10) and will be older and middle-aged adults (55+). Clients will be identified by senior center staff trained in SMART-MH strategies. Investigators will offer additional training to staff of all centers on SMART-MH outreach, depression screening, and treatment engagement. Investigators will train and provide weekly supervision to 2 or more LCSWs per center of the two centers assigned to Engage-M. Investigators will not offer training or supervision to senior center staff leading the groups of W-MH but will provide oversight so that clients receive mental health referrals and are encouraged to attend weekly Wellness group meetings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engage-M (Experimental): Participants will meet individually with a therapist once before beginning weekly group sessions for eight weeks. Each weekly session will last approximately 50 minutes. Study investigators have trained Engage-M therapists to provide participants with a group therapy approach called Engage-M. During the weekly therapy sessions, therapists will encourage participants to engage in physical and social activities that you find pleasurable or rewarding.
  Interventions: Behavioral: Engage-M
- Wellness in Mind and Body (W-MH) (Active Comparator): Participants will meet with a therapist for group therapy once a week for eight weeks. Each weekly session will last approximately 50 minutes. During these weekly sessions, the therapist will educate participants about health and mental health.
  Interventions: Behavioral: Wellness in Mind and Body

INTERVENTIONS:
Behavioral: Engage-M — Engage is a stepped care psychotherapy based on what is known about how older adults respond to depression interventions. Stepped care is a model of treatment that starts with the minimum effective therapeutic techniques first, and then based on how well people respond to treatment, additional therapeutic techniques are added until people are recovered from their depression.
  Arms: Engage-M
Behavioral: Wellness in Mind and Body — An active intervention focusing on psychoeducation and de-stigmatization of health and mental health conditions. These sessions are commonly part of senior centers programs. W-MH will offer mental health referral to a clinic or primary care physician as part of senior center procedures for clients with positive PHQ-9s.
  Other Names: W-MH
  Arms: Wellness in Mind and Body (W-MH)

SUMMARY:
The purpose of this study is to test the feasibility of two types of group therapy sessions. The research is being done because the researchers are trying to learn if these approaches could be used by therapist in the community social service agencies to treat older adults with depression. There are two study groups. One group is a form of group therapy called "Engage-M", which encourages subjects to engage in physical and social activities that they find pleasurable or rewarding. One group is another form of group therapy called, "Wellness in Mind and Body", which focuses on education and de-stigmatization of health and mental health conditions.

DETAILED DESCRIPTION:
In response to the large numbers of senior center clients who suffer from untreated depression, we have partnered with the NYC Department for the Aging (DFTA) to develop SMART-MH, a community care model that can be embedded in senior centers to improve recognition, referral, and adherence to depression treatment. The investigators also developed and tested Engage, a stepped-care therapy streamlined to use "reward exposure" as its principal intervention based on the assumption that dysfunction of the reward networks is central to the pathogenesis of depression. With senior center partners and a mobile technology team, the investigators redesigned Engage-M so that it can be used in a group format by licensed clinical social workers (LCSWs) of Senior Centers. Mobile technology provides probes for client adherence and offers to therapists easy to review summary records of mood, activity, and social interaction that can be used to target their sessions. The investigators have integrated SMART-MH and Engage-M into a comprehensive community care model "Reaching and Engaging Depressed Senior Center Clients" (REDS).

The specific aims of this developmental project are to: 1. Finalize the REDS protocol and assess feasibility of training; 2. Prepare an Operations' Manual; 3. Examine reach, feasibility, and acceptability of REDS; 4. Examine engagement of behavioral targets and preliminary effectiveness; and 5. Collect information on REDS cost, barriers to implementation, and potential savings in health care utilization.

The investigators will randomly assign four senior centers to offer either Engage-M (N=40), the treatment offered by REDS (1 individual and 8 weekly group sessions) or 8 group sessions "Wellness in Mind and Body" plus mental health referral (W-MH; N=20). The participants will have clinically significant depressive symptoms (PHQ-9>10) and will be older and middle-aged adults (55+); 12.6% of the NYC senior center clients are aged 55-65 years. Clients will be identified by senior center staff trained in SMART-MH strategies. The investigators will offer additional training to staff of all centers on SMART-MH outreach, depression screening, and treatment engagement. The investigators will train and provide weekly supervision to 2 or more LCSWs per center of the two centers assigned to Engage-M. The investigators will not offer training or supervision to senior center staff leading the groups of W-MH but will provide oversight so that clients receive mental health referrals and are encouraged to attend weekly Wellness group meetings.

ELIGIBILITY:
Inclusion Criteria:

* 55 years+
* PHQ-9≥10
* English or Spanish speaking
* MMSE ≥ 24
* Capacity to provide written consent for both research assessment and the Engage-M intervention.

Exclusion Criteria:

* Current active suicidal ideation defined by MADRS Suicide Item ≥ 4 (Probably better off dead. Suicidal thoughts are common, and suicide is considered as a possible solution, but without specific plans or intention).
* Presence of psychiatric diagnoses other than unipolar, non-psychotic major depression pr generalized anxiety disorder by SCID-V.
* Severe or life-threatening medical illness (e.g. end-stage organ failure).

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Alexopoulos, MD, Study Director — Weill Medical College of Cornell University; Patricia Marino, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The Center will share its data via the NIMH Data Archive (NDA). The resource sharing plan is formulated in accordance with the NDA Data Sharing Terms and Conditions. Further, the Center will use NDA technologies to submit data in accordance with the NDA Data Sharing Terms and Conditions.
  The investigators will comply with NIMH's procedures for data deposition into NDCT, and will let NDCT policies dictate the timetable upon which and avenues through which others will be allowed to access those data. Investigators will make the dataset available to other researchers after the main results have been published. Investigators will de-identify the data in the final datasets prior to release for sharing. To ensure data and participant security, investigators will make the data available to users only under a data-sharing agreement.
Time Frame: Per NIMH guidelines.
Access Criteria: All users will first provide to the ALACRITY Center and the co-Investigators with a proposal of hypotheses, variables needed to test these hypotheses, and plans for dissemination of findings. All users will indicate in a signed document: (1) a commitment to using the data only for research purposes; (2) a plan for securing the data; (3) an agreement to either destroying or returning the data once analyses are completed; and (4) an agreement to not share data with other users and to direct all such requests to The ALACRITY Center.
  Findings will be reported in scientific meetings and publications promptly. Consistent with NIH policy, publications will be deposited at PubMed Central. The data from this research will be made available for integration with other datasets of the ALACRITY Center.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engage-M | Wellness in Mind and Body (W-MH)
Started | 24 | 15
Completed | 24 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engage-M | Wellness in Mind and Body (W-MH) | Total
Number analyzed (Participants) | 24 | 15 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.88 (6.91) | 73.60 (7.40) | 72.54 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 35
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 20 | 15 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 14 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 24 | 15 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinically Significant Depressive Symptoms (MADRS)
Description: In both conditions, the change in clinically significant depressive symptoms as measured on the Montgomery Asberg Depression Rating Scale (MADRS). The scale captures the severity of ten common symptoms of depression. The combined score yields a value between 0-60. Higher scores indicate more severe depression, which benchmarks as follows: 0 to 6: normal/symptoms absent; 7 to 19: mild depression; 20 to 34: moderate depression; >34: severe depression.
Time Frame: These measures are assessed at baseline, six week, nine week and twelve weeks after study enrollment-during the study-to document change in depressive symptoms.
Population: Engage-M: Two participants completed only their baseline assessment. Additionally, two participants did not attend their Week-6 assessment, and one participant did not attend their Week-9 assessment.
  Wellness in Mind and Body (W-MH): One participant completed only their baseline assessment. Additionally, one participant did not attend their Week-6 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage-M | Wellness in Mind and Body (W-MH)
Number analyzed (Participants) | 24 | 15
score on a scale
  Baseline | 21.21 (5.38) | 21 (3.85)
  Week 6: number analyzed (Participants) | 20 | 13
  Week 6 | 18.5 (5.88) | 15.77 (6.18)
  Week 9: number analyzed (Participants) | 21 | 14
  Week 9 | 15.86 (6.78) | 15.86 (4.38)
  Week 12: number analyzed (Participants) | 22 | 14
  Week 12 | 15.36 (5.69) | 13.21 (6.25)
Statistical Analysis 1: Comparison: Engage-M vs Wellness in Mind and Body (W-MH); Week 12; Test type: Superiority; p = 0.31, t-test, 2 sided; Mean Difference (Final Values) = 2.15, 95% CI 2-sided [-2.09 to 6.39]

2. Secondary Outcome: Change in Assessment of Quality of Life (WHO-QOL)
Description: In both conditions, change in assessment of quality of life is measured by the World Health Organization Quality of Life (WHOQOL) scale. This scale measures quality of life across four domains: 1) Physical Health 2) Psychological 3) Social relationships and 4) Environment. A higher score in any domain indicates a better outcome, and min/max values for each domain are as follows: 1) 7-35 2) 6-30 3) 3-15 4) 8-40.
Time Frame: These measures are assessed at baseline, six week, nine week and twelve weeks after study enrollment-during the study-to document change in assessment of quality of life.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage-M | Wellness in Mind and Body (W-MH)
Number analyzed (Participants) | 24 | 15
score on a scale
  Baseline - Domain 1 | 22.14 (4.10) | 20.87 (3.23)
  Baseline - Domain 2 | 17.81 (3.43) | 17.50 (3.03)
  Baseline - Domain 3 | 8.30 (2.62) | 9.36 (1.43)
  Baseline - Domain 4 | 29.00 (4.01) | 30.80 (3.76)
  Week 6 - Domain 1: number analyzed (Participants) | 20 | 13
  Week 6 - Domain 1 | 22.16 (3.78) | 21.00 (3.57)
  Week 6 - Domain 2: number analyzed (Participants) | 20 | 13
  Week 6 - Domain 2 | 18.00 (3.35) | 18.83 (2.52)
  Week 6 - Domain 3: number analyzed (Participants) | 20 | 13
  Week 6 - Domain 3 | 8.92 (2.14) | 9.00 (2.49)
  Week 6 - Domain 4: number analyzed (Participants) | 20 | 13
  Week 6 - Domain 4 | 31.42 (4.34) | 30.25 (5.05)
  Week 9 - Domain 1: number analyzed (Participants) | 21 | 14
  Week 9 - Domain 1 | 22.67 (2.37) | 22.08 (4.42)
  Week 9 - Domain 2: number analyzed (Participants) | 21 | 14
  Week 9 - Domain 2 | 18.19 (3.28) | 19.08 (4.41)
  Week 9 - Domain 3: number analyzed (Participants) | 21 | 14
  Week 9 - Domain 3 | 9.08 (2.68) | 10.00 (1.49)
  Week 9 - Domain 4: number analyzed (Participants) | 21 | 14
  Week 9 - Domain 4 | 31.43 (4.04) | 29.69 (4.52)
  Week 12 - Domain 1: number analyzed (Participants) | 22 | 14
  Week 12 - Domain 1 | 20.68 (4.19) | 22.15 (3.76)
  Week 12 - Domain 2: number analyzed (Participants) | 22 | 14
  Week 12 - Domain 2 | 17.59 (3.84) | 18.46 (3.67)
  Week 12 - Domain 3: number analyzed (Participants) | 22 | 14
  Week 12 - Domain 3 | 8.69 (2.55) | 10.27 (1.27)
  Week 12 - Domain 4: number analyzed (Participants) | 22 | 14
  Week 12 - Domain 4 | 30.18 (4.69) | 30.23 (5.33)
Statistical Analysis 1: Comparison: Engage-M vs Wellness in Mind and Body (W-MH); Domain #1, Week 12; Test type: Superiority; p = 0.28, t-test, 2 sided; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-4.22 to 1.28]
Statistical Analysis 2: Comparison: Engage-M vs Wellness in Mind and Body (W-MH); Domain #2, Week 12; Test type: Superiority; p = 0.50, t-test, 2 sided; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-3.48 to 1.74]
Statistical Analysis 3: Comparison: Engage-M vs Wellness in Mind and Body (W-MH); Domain #3, Week 12; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-2.88 to -0.28]
Statistical Analysis 4: Comparison: Engage-M vs Wellness in Mind and Body (W-MH); Domain 4, Week 12; Test type: Superiority; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-3.63 to 3.53]

3. Other Pre Specified Outcome: Change in Satisfaction With Study Intervention (CSQ)
Description: Client satisfaction with study intervention as measured by the Client Satisfaction Questionnaire (CSQ) in both treatments. The questionnaire comprises three questions, rated on a scale of 1-4. A higher score indicates a greater degree of client satisfaction.
  1. To what extent has the study therapist met your needs? 4=Almost all of my needs have been met 3=Most of my needs have been met 2=Some of my needs have been met 1=None of my needs have been met
  2. In an overall sense, how satisfied are you with the services that you have received? 4=Very satisfied 3=Mostly satisfied 2=Indifferent or mildly dissatisfied 1=Quite dissatisfied
  3. If you were to seek help again, would you come back to the study therapist you are currently seeing? 4=Yes, definitely 3=Yes, I think so 2=No, I don't think so 1=No, definitely not
Time Frame: Assessed after REDS sessions completed at six, nine, and twelve weeks after study enrollment.
Population: Engage-M: Two participants did not attend their Week-6 assessment, and one participant did not attend their Week-9 assessment.
  Wellness in Mind and Body (W-MH): One participant did not attend their Week-6 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage-M | Wellness in Mind and Body (W-MH)
Number analyzed (Participants) | 22 | 14
score on a scale
  Week 6 - #1: number analyzed (Participants) | 20 | 13
  Week 6 - #1 | 2.80 (1.06) | 2.23 (0.73)
  Week 6 - #2: number analyzed (Participants) | 20 | 13
  Week 6 - #2 | 3.35 (0.88) | 2.77 (0.93)
  Week 6 - #3: number analyzed (Participants) | 20 | 13
  Week 6 - #3 | 3.50 (0.76) | 3.69 (0.48)
  Week 9 - #1: number analyzed (Participants) | 21 | 14
  Week 9 - #1 | 3.00 (1.00) | 2.43 (0.65)
  Week 9 - #2: number analyzed (Participants) | 21 | 14
  Week 9 - #2 | 3.57 (0.75) | 3.14 (0.77)
  Week 9 - #3: number analyzed (Participants) | 21 | 14
  Week 9 - #3 | 3.70 (0.57) | 3.50 (0.76)
  Week 12 - #1 | 2.68 (0.95) | 2.71 (0.83)
  Week 12 - #2 | 3.18 (0.80) | 3.36 (0.63)
  Week 12 - #3 | 3.68 (0.72) | 3.50 (0.76)
Statistical Analysis 1: Comparison: Engage-M vs Wellness in Mind and Body (W-MH); Domain #1, Week 12; Test type: Superiority; p = 0.92, t-test, 2 sided; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.64 to 0.58]
Statistical Analysis 2: Comparison: Engage-M vs Wellness in Mind and Body (W-MH); Domain #2, Week 12; Test type: Superiority; p = 0.48, t-test, 2 sided; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.69 to 0.33]
Statistical Analysis 3: Comparison: Engage-M vs Wellness in Mind and Body (W-MH); Test type: Superiority; p = 0.48, t-test, 2 sided; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.33 to 0.69]

ADVERSE EVENTS:
Time Frame: Each participant was monitored for adverse events for twelve weeks after the completion of their baseline assessment.
Arm/Group | Engage-M | Wellness in Mind and Body (W-MH)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/15
Other Adverse Events (participants affected / at risk) | 0/24 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT03246789/Prot_000.pdf